CLINICAL TRIAL: NCT03735238
Title: Implementing the Decision-Aid for Lupus (IDEAL Strategy)
Acronym: IDEAL
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jasvinder A Singh, Faculty, University of Alabama at Birmingham
Other Study IDs: 300002272; CE-1304-6631 (Other Grant/Funding Number: PATIENT-CENTERED OUTCOMES RESEARCH INSTITUTE (PCORI))
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; decision making; implementation; SLE; decision-aid; decision conflict
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lupus Patients: All adult lupus patients, regardless of if they are having an active flare
  Interventions: Other: SMILE Computerized Decision-Aid

INTERVENTIONS:
Other: SMILE Computerized Decision-Aid — SMILE is a computerized decision-aid designed to give lupus patients information about lupus, treatments for lupus available to them, as well as side effects. This will be administered at every lupus clinic session. Every patient will see the SMILE Computerized Decision-Aid at their index baseline clinic visit.
  Other Names: SMILE; Decision-Aid; DA

SUMMARY:
The study will attempt to put into practice a shared decision making (SDM) strategy, using an individualized, computerized decision- aid (DA) for Systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
The proposed study will evaluate methods to implement a shared decision making strategy, using an individualized, computerized decision- aid (DA). The investigators will test the effectiveness of this implementation with 3 strategies in 15 clinics. Formative evaluation strategies will be used to assess needs at each clinic, with key clinic informants participating in semi-structured interviews. The study will enroll patient participants across all 16 sites, who will review the decision aid and be asked a feasibility and acceptability assessment. At the conclusion of the study, key clinic informants, as well as selected patient participants will participate in semi-structured interviews to assess the effectiveness in implementing the DA in the clinic setting.

ELIGIBILITY:
Patient Inclusion Criteria:

* Adults with a diagnosis of Systemic Lupus Erythematosus (SLE) by a rheumatologist

Patient Exclusion Criteria:

* No diagnosis of lupus, not English or Spanish speaking, visually impaired, altered mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from lupus clinics at 15 sites throughout the country.
Sampling Method: Non-Probability Sample
Enrollment: 1895 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder A Singh, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh JA, Hearld LR, Eisen S, Chatham WW, Narain S, Annapureddy N, Kamen DL, Trotter K, Majithia V, Ching CL, Aouhab Z, Venuturupalli S, Wallace DJ, Ramsey-Goldman R, Kim AHJ, McMahon M, Lim SS, Bhairavarasu K, Meara A, Kalunian K, Beasley M. Patient outcomes from implementing a shared decision-making aid for systemic lupus erythematosus: a prospective implementation study. Lancet Rheumatol. 2025 Sep 17:S2665-9913(25)00130-4. doi: 10.1016/S2665-9913(25)00130-4. Online ahead of print. PMID 40975111
- [Derived] Singh JA, Beasley TM. Association of Patient Resilience With Patient-Reported Physical and Mental/Emotional Quality of Life in Systemic Lupus Erythematosus. J Rheumatol. 2025 Dec 1;52(12):1263-1273. doi: 10.3899/jrheum.2025-0396. PMID 40953958
- [Derived] Singh JA, Hearld LR, Eisen S, Chatham WW, Narain S, Annapureddy N, Kamen DL, Trotter K, Majithia V, Lee Ching C, Aouhab Z, Venuturupalli S, Wallace DJ, Ramsey-Goldman R, Kim A, McMahon M, Sam Lim S, Bhairavarasu K, Meara A, Kalunian K, Beasley TM; Implementing DEcision-Aid for Lupus in clinics (IDEAL) Consortium. Implementation outcomes of a patient decision-aid in a diverse population with systemic lupus erythematosus in 15 US rheumatology clinics. Rheumatology (Oxford). 2025 Aug 1;64(8):4631-4640. doi: 10.1093/rheumatology/keaf205. PMID 40221856
- [Derived] Blanchard EE, Hall AG, Gore E, Jami PY, Karabukayeva A, Hearld LR, Gontarz S, Singh JA. Barriers to and facilitators of sustaining a systemic lupus erythematosus (SLE) patient decision aid in regular rheumatology outpatient care in the USA. Rheumatology (Oxford). 2025 Jun 1;64(6):3580-3586. doi: 10.1093/rheumatology/keaf043. PMID 39873723
- [Derived] Singh JA, Hearld LR, Hall AG, Beasley TM. Implementing the DEcision-Aid for Lupus (IDEAL): study protocol of a multi-site implementation trial with observational, case study design : Implementing the DEcision-Aid for Lupus. Implement Sci Commun. 2021 Mar 11;2(1):30. doi: 10.1186/s43058-021-00118-9. PMID 33706813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 15 participating sites were asked to enroll a minimum number of SLE patient participants at the site (n=28/site), and to continue enrolling once the threshold was met. The clinic personnel were not enrolled.
Groups:
- Lupus Patients: All lupus patients, regardless of if they are having an active flare, participated. There was no randomly assigned arms or conditions.
Period: Overall Study
Arm/Group | Lupus Patients
Started | 1895
Completed | 1866
Not Completed | 29
Not completed — Did not want to participate in research | 3
Not completed — Time constraints, patient preference or percieved burden of survey completion | 26

BASELINE CHARACTERISTICS:
Groups:
- Lupus Patients: All lupus patients, regardless of if they are having an active flare.
Arm/Group | Lupus Patients
Number analyzed (Participants) | 1855
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data = 6
  years
    number analyzed (Participants) | 1849
    (all) | 44.68 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1731
  Male | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data = 23
  Participants
    Race: number analyzed (Participants) | 1832
    Race: Asian | 80
    Race: African American | 827
    Race: Hispanic | 149
    Race: Other/Mixed | 22
    Race: White | 754
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data = 21
  Participants
    Ethnicity: number analyzed (Participants) | 1834
    Ethnicity: Hispanic or Latino | 149
    Ethnicity: Not Hispanic or Latino | 1685
Insurance Payer Type [Count of Participants; unit: Participants] — Population: Missing data = 405 (Insurance payer type question was added much later after the start of the study, based on stakeholder feedback, therefore missingness is higher for this variable)
  Participants
    number analyzed (Participants) | 1450
    Commercial/Private | 655
    Medicare | 340
    Medicaid | 221
    Other | 234
Education level [Count of Participants; unit: Participants] — Population: Missing data = 849 (Education level question was added much later after the start of the study, based on stakeholder feedback, therefore missingness is higher for this variable)
  Participants
    number analyzed (Participants) | 1006
    Less than HS | 27
    HS degree or GED | 152
    Greater than HS | 827
Marital status [Count of Participants; unit: Participants] — Population: Missing data = 849 (Marital status question was added much later after the start of the study, based on stakeholder feedback, therefore missingness is higher for this variable)
  Participants
    number analyzed (Participants) | 1006
    Married | 443
    Separated | 19
    Divorced | 87
    Single | 372
    Living with partner | 45
    Widowed | 33
    Other | 7
Residence [Count of Participants; unit: Participants] — Population: Missing data = 849 (Residence question was added much later after the start of the study, based on stakeholder feedback, therefore missingness is higher for this variable)
  Participants
    number analyzed (Participants) | 1006
    Urban | 305
    Suburban | 483
    Rural | 218

OUTCOME MEASURES:

1. Primary Outcome: Penetration/Reach: Number of Eligible Participants at Each Clinical Site Who Enrolled Divided by the Number of Eligible Participants at Each Clinical Site, Expressed as Overall Percent
Description: Reach/penetration was measured by calculating a ratio of patients who were enrolled in the implementation project (# of patients who viewed the SLE PtDA) divided by the number of Eligible Participants at Each Clinical Site identified using the electronic medical record (EMR) in the respective clinic (# of eligible patients). The number of eligible patients was based on the average number of patients with a diagnosis of lupus seen in each clinic over the study period (2019-2023).
Time Frame: 24 months
Population: Reach/penetration = # of patients viewed DA / # of eligible patients
Measure: Number; unit: Participants
Groups:
- Loyola University, Chicago: Penetration of DA at Loyola University, Chicago
- University of Alabama at Birmingham (UAB), Birmingham: Penetration of DA at University of Alabama at Birmingham, Birmingham, Alabama
- Vanderbilt University, Nashville: Penetration of DA at Vanderbilt University, Nashville, Tennessee
- University of Chicago, Chicago: Penetration of DA at the University of Chicago, Chicago (UChicago), Illinois
- University of Mississippi Medical Center (UMMC), Jackson: Penetration of DA at the University of Mississippi Medical center, Jackson, Mississippi
- Cedars Cedars-Sinai Medical Center, Los Angeles: Penetration of DA at Cedars-Sinai Medical Center, Los Angeles, California
- Baylor College of Medicine, Houston: Penetration of DA at the Baylor College of Medicine, Houston, Texas
- Northwestern University, Chicago: Penetration of DA at the Northwestern University, Chicago, Illinois
- Emory University, Atlanta: Penetration of DA at the Emory University, Atlanta, Georgia
- Medical University of South Carolina (MUSC), Charleston: Penetration of DA at the Medical University of South Carolina (MUSC), Charleston, SC
- Northwell Health, New York: Penetration of DA at the Northwell Health, New York, New York
- University of California (UCLA), Los Angeles: Penetration of DA at the University of California (UCLA), Los Angeles, California
- Ohio State University (OSU), Columbus: Penetration of DA at the Ohio State University (OSU), Columbus, Ohio
- University of California at San Diego (UCSD), San Diego, CA: Penetration of DA at the University of California at San Diego (UCSD), San Diego, CA
- Washington University, St. Louis: Penetration of DA at the Washington University, St. Louis, Missouri
Arm/Group | Loyola University, Chicago | University of Alabama at Birmingham (UAB), Birmingham | Vanderbilt University, Nashville | University of Chicago, Chicago | University of Mississippi Medical Center (UMMC), Jackson | Cedars Cedars-Sinai Medical Center, Los Angeles | Baylor College of Medicine, Houston | Northwestern University, Chicago | Emory University, Atlanta | Medical University of South Carolina (MUSC), Charleston | Northwell Health, New York | University of California (UCLA), Los Angeles | Ohio State University (OSU), Columbus | University of California at San Diego (UCSD), San Diego, CA | Washington University, St. Louis
Number analyzed (Participants) | 200 | 1612 | 447 | 522 | 463 | 512 | 389 | 500 | 818 | 1388 | 2087 | 1292 | 666 | 850 | 1148
Participants | 96 | 725 | 121 | 104 | 105 | 88 | 63 | 79 | 73 | 102 | 124 | 69 | 37 | 28 | 81
Statistical Analysis 1: Comparison: Loyola University, Chicago vs University of Alabama at Birmingham (UAB), Birmingham vs Vanderbilt University, Nashville vs University of Chicago, Chicago vs University of Mississippi Medical Center (UMMC), Jackson vs Cedars Cedars-Sinai Medical Center, Los Angeles vs Baylor College of Medicine, Houston vs Northwestern University, Chicago vs Emory University, Atlanta vs Medical University of South Carolina (MUSC), Charleston vs Northwell Health, New York vs University of California (UCLA), Los Angeles vs Ohio State University (OSU), Columbus vs University of California at San Diego (UCSD), San Diego, CA vs Washington University, St. Louis; This is a single arm implementation trial with no comparison group. This outcome represents the reach/penetration of the implementation at each site over the trial duration. We did not perform power calculation. There was no null hypothesis stated. Our aim was to enroll at least 28 patients per site in this implementation trial during regular outpatient rheumatology clinic visits. No statistical test was performed for this outcome; Test type: Other — Not applicable. No statistical test was performed for this outcome; Our aim was to enroll at least 28 patients per site in this implementation trial during regular outpatient rheumatology clinic visits. No statistical test was performed for this outcome

2. Secondary Outcome: Perceived Acceptability of Intervention Measure (AIM) by Clinic Personnel for the SLE Patient Decision-aid
Description: Clinic personnel's perception of the acceptability of the SLE Patient decision-aid (PtDA), measured using a validated scale with four (4) items with responses ranging from 1 ("completely disagree") to 5 ("completely agree"). The four items will be averaged to create one composite mean scale score (range 1-5), where higher scores reflect perceptions of greater acceptability (i.e., better outcome).
Time Frame: 24 months
Population: The main study flow diagram is for the patient participants who were invited to view the SLE PtDA. We also evaluated clinic personnel reported outcomes, which are provided for outcomes #2-6, including this outcome. As expected, the denominator for the clinic personnel outcomes is different from that for the patient participants. In summary, our implementation study had separate aims focused on patient-reported effectiveness outcomes, and clinic personnel reported implementation outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Groups:
- 4-months Post-implementation: Clinic Personnel's acceptability of DA 4-months post-implementation
- 12-months Post-implementation: Clinic Personnel's acceptability of DA12-months post-implementation
- 24-months Post-implementation: Clinic Personnel's acceptability of DA 24-months post-implementation
Arm/Group | 4-months Post-implementation | 12-months Post-implementation | 24-months Post-implementation
Number analyzed (Participants) | 97 | 82 | 70
score on a scale (range 1-5) | 3.53 (0.83) | 3.84 (0.80) | 3.63 (0.79)

3. Secondary Outcome: Perceived DA Implementation Success by Clinic Personnel for the SLE Patient Decision-aid
Description: Clinic personnel's perception of the implementation success of the SLE Patient decision-aid (PtDA), measured using a validated scale with three (3) items with responses ranging from 1 ("Disagree") to 5 ("Agree"). These three items will be averaged to create one composite mean scale score (range 1-5), where higher scores reflect perceptions of greater implementation success (i.e., better outcome).
Time Frame: 24 months
Population: The main study flow diagram is for the patient participants. We also evaluated clinic personnel reported outcomes in this study, which are provided for outcomes #2-6, including this outcome. The denominator for the clinic personnel is different from those of the patient participants, as expected.
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Groups:
- 4-months Post-implementation: Clinic personnel's perceived implementation of success of the Decision Aid (DA) 4-months post-implementation
- 12-months Post-implementation: Clinic personnel's perceived implementation of success of the Decision Aid (DA) 12-months post-implementation
- 24-months Post-implementation: Clinic personnel's perceived implementation of success of the Decision Aid (DA) 24-months post-implementation
Arm/Group | 4-months Post-implementation | 12-months Post-implementation | 24-months Post-implementation
Number analyzed (Participants) | 97 | 82 | 70
score on a scale (range 1-5) | 3.41 (0.73) | 3.54 (0.70) | 3.47 (0.91)

4. Secondary Outcome: Perceived DA Permanence by Clinic Personnel for the SLE Patient Decision-aid
Description: Clinic personnel's perception of the permanence of the SLE Patient decision-aid (PtDA), measured using one validated item that is scored ranging from 1 ("Not at all permanent") to 5 ("Extremely permanent"). This item will be examined by itself, where higher scores indicate perceptions of greater permanence of the decision-aid in the clinic (i.e., better outcome).
Time Frame: 24 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Groups:
- 4-months Post-implementation: Clinic personnel's perceived Decision Aid (DA) permanence of the decision-aid 4-months post-implementation
- 12-months Post-implementation: Clinic personnel's perceived Decision Aid (DA) permanence of the decision-aid 12-months post-implementation
- 24-months Post-implementation: Clinic personnel's perceived Decision Aid (DA) permanence of the decision-aid 24-months post-implementation
Arm/Group | 4-months Post-implementation | 12-months Post-implementation | 24-months Post-implementation
Number analyzed (Participants) | 99 | 79 | 70
score on a scale (range 1-5) | 3.22 (0.74) | 3.02 (0.96) | 3.11 (1.03)

5. Secondary Outcome: Perceived Intervention Appropriateness Measure (IAM) by Clinic Personnel for the SLE Patient Decision-aid
Description: Clinic personnel's perception of the appropriateness of the SLE Patient decision-aid (PtDA), measured using a validated scale with four (4) items with responses ranging from 1 ("completely disagree") to 5 ("completely agree"). The four items will be averaged to create one composite mean scale score (range 1-5), where higher scores reflect perceptions of greater appropriateness (i.e., better outcome).
Time Frame: 24 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Groups:
- 4-months Post-implementation: Clinic personnel's perceived Intervention Appropriateness Measure (IAM) for Decision Aid (DA) 4-months post-implementation
- 12-months Post-implementation: Clinic personnel's perceived Intervention Appropriateness Measure (IAM) for Decision Aid (DA)12-months Post-implementation
- 24-months Post-implementation: Clinic personnel's perceived Intervention Appropriateness Measure (IAM) for Decision Aid (DA) 24-months post-implementation
Arm/Group | 4-months Post-implementation | 12-months Post-implementation | 24-months Post-implementation
Number analyzed (Participants) | 98 | 79 | 69
score on a scale (range 1-5) | 3.43 (0.86) | 3.76 (0.74) | 3.64 (0.85)

6. Secondary Outcome: Perceived Feasibility of Intervention Measure (FIM) by Clinic Personnel for the SLE Patient Decision-aid
Description: Clinic personnel's perception of the feasibility of the SLE Patient decision-aid (PtDA), measured using a validated scale with four (4) items with responses ranging from 1 ("completely disagree") to 5 ("completely agree"). The four items will be averaged to create one composite mean scale score (range 1-5), where higher scores reflect perceptions of greater feasibility (i.e., better outcome).
Time Frame: 24 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Groups:
- 4-months Post-implementation: Clinic personnel's perceived Feasibility of Intervention Measure (FIM) for Decision Aid (DA) 4-months post-implementation
- 12-months Post-implementation: Clinic personnel's perceived Feasibility of Intervention Measure (FIM) for Decision Aid (DA) 12-months post-implementation
- 24-months Post-implementation: Clinic personnel's perceived Feasibility of Intervention Measure (FIM) for Decision Aid (DA) 24-months post-implementation
Arm/Group | 4-months Post-implementation | 12-months Post-implementation | 24-months Post-implementation
Number analyzed (Participants) | 100 | 79 | 70
score on a scale (range 1-5) | 3.44 (0.71) | 3.61 (0.75) | 3.53 (0.81)

7. Secondary Outcome: Patient Decisional Conflict Scale Related to Medication Treatment Decision-making for SLE Medications Including the Immunosuppressive Medications and Biologics After Viewing the SLE Patient Decision-aid
Description: Decisional conflict was measured using the low literacy version of the Decisional Conflict Scale (DCS), a well-validated self-administered instrument, after viewing the SLE Patient decision-aid (PtDA). The low literacy version has 10 items with 3 response categories: yes, unsure, and no. Four subscale scores consisting of uncertainty about choice, feeling informed, values clarity, and feeling supported in decision-making were also calculated. DCS (and subscale) scores range from 0 (best) to 100 (worst) and scores >= 25 are consistent with clinically significant residual decisional conflict
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale (DCS; 0-100)
Groups:
- Baseline Visit: Patient viewing of Lupus Decision-aid (DA) at baseline visit
- 3-Month Visit: Patient viewing of Lupus Decision-aid (DA) at 3 Month visit
- 6 Month Visit: Patient viewing of Lupus Decision-aid (DA) at 6 Month visit
Arm/Group | Baseline Visit | 3-Month Visit | 6 Month Visit
Number analyzed (Participants) | 1849 | 1211 | 1255
score on a scale (DCS; 0-100) | 19.48 (23.78) | 21.77 (25.70) | 20.23 (24.67)

8. Secondary Outcome: Patient-reported Interpersonal Processes of Care for Patient-Physician Communication After Viewing the SLE Patient Decision-aid
Description: The Interpersonal Processes of Care short form (IPC-SF) is a patient-reported, 18-item validated patient-reported patient-physician communication and care processes measure, assessed after viewing the SLE Patient decision-aid (PtDA). Scores range from 18 to 90, with higher scores indicating better patient-physician communication ± care.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale (IPC; 18-90)
Arm/Group | Baseline Visit | 3-Month Visit | 6 Month Visit
Number analyzed (Participants) | 1844 | 1207 | 1255
score on a scale (IPC; 18-90) | 82.19 (9.28) | 81.88 (9.84) | 82.34 (9.36)

9. Secondary Outcome: Patient Satisfaction for SLE Patient Decision-aid
Description: Patient satisfaction with the ease of the use of the SLE Patient Decision-aid (PtDA) measured using a validated single item scale scored on an ordinal scale from (strongly disagree =1) to (strongly agree = 5). This item will be examined by itself, where higher scores indicate greater patient satisfaction with the decision aid (i.e., better outcome). This is a single item scale, and there are no subscales. It was adapted from another study that assessed satisfaction with iPad or interactive voice response.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-5)
Arm/Group | Baseline Visit | 3-Month Visit | 6 Month Visit
Number analyzed (Participants) | 1839 | 1197 | 1237
score on a scale (range 1-5) | 4.41 (1.08) | 4.44 (0.87) | 4.44 (0.85)

10. Secondary Outcome: Patient Time for Reviewing SLE Patient Decision-aid
Description: The SLE Patient Decision-aid (PtDA) review times was expressed in minutes as patient-reported; this was supplemented by study coordinator's record of patient DA review time in-clinic prior to addition of this question. This patient self-reported question was added at the onset of the COVID-19 pandemic, where shelter-in-place orders led to stopping of in-person outpatient visits and all vists were converted to virtual visits using the phone or the video (Telemedicine).
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Baseline Visit | 3-Month Visit | 6 Month Visit
Number analyzed (Participants) | 755 | 477 | 509
Minutes | 23 (16.18) | 22.44 (13.44) | 21.63 (14.81)

11. Secondary Outcome: Patient Preparation for Decision Making Assessed After Viewing the SLE Patient Decision-aid
Description: Patient perception of the effect of the decision-aid on preparing the patient for decision making measured using the Patient Preparation for Decision Making (PDM) , a validated scale consisting of 10 questions scored on an ordinal scale from (not at all =1) to (a great deal = 5. Score ranged 0-100, 100 representing the highest preparation for decision-making. This was assessed after viewing the SLE Patient decision-aid (PtDA).
Time Frame: Baseline visit after viewing the SLE Patient Decision-Aid (PtDA)
Population: All SLE Patients who viewed the SLE PtDA patients, regardless of if they are having an active flare, and responded to this part of the patient survey
Measure: Mean (Standard Deviation); unit: score on a scale (PDM; 0-100)
Groups:
- SLE Patients Who Viewed the SLE PtDA: All SLE Patients who viewed the SLE PtDA patients, regardless of if they are having an active flare, and responded to this part of the patient survey
Arm/Group | SLE Patients Who Viewed the SLE PtDA
Number analyzed (Participants) | 1827
score on a scale (PDM; 0-100) | 74.44 (23.76)

12. Secondary Outcome: Patient Acceptability of the SLE Patient Decision-Aid
Description: The patient acceptability survey is for the assessment of patient acceptability of the SLE Patient Decision-Aid (PtDA). Each question was rated from Poor (1) to Excellent (4). Total score ranged 1-4. DA acceptability refers to rating regarding the comprehensibility of component of the decision-aid, its length, pace, amount of the information, and the balance in presentation of the information about the options available and the overall suitability for decision making.
Time Frame: Baseline visit after viewing the SLE PtDA
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale (range:1-4)
Arm/Group | Lupus Patients
Number analyzed (Participants) | 1858
score on a scale (range:1-4) | 3.26 (0.63)

13. Secondary Outcome: Patient Feasibility of the SLE Patient Decision-Aid
Description: The feasibility of the study survey completion and the administration of the lupus decision aid in the busy clinic were assessed with a self-administered patient questionnaire consisting of 4 questions, 2 questions for each, the survey and for the process of viewing ± administering the lupus DA in the busy clinic. Responses ranged from strongly disagree (=1) to strongly agree (=5). Higher scores indicate higher feasibility of the survey and of the SLE Patient Decision-Aid (PtDA) administration respectively.
Time Frame: Baseline visit after viewing the SLE PtDA
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale (range:1-4)
Arm/Group | Lupus Patients
Number analyzed (Participants) | 1822
score on a scale (range:1-4) | 4.33 (0.77)

14. Secondary Outcome: Number of Participants Who Perceived the SLE Patient Decision-Aid to be Useful
Description: Patient perception of the SLE Patient Decision-Aid (PtDA) usefulness was aimed at assessing whether people would consider the the SLE PtDA to be useful at present and when they would think back to the time, they had made decisions about lupus treatments in the past (question 1), and whether the information contained in the lupus DA were adequate (question 2). It measured patient response of Yes vs. no to two simple questions. The tool is not yet a validated assessment but was based on our debriefing of lupus patients in the previous randomized study of lupus decision-aid.
Time Frame: Baseline visit after viewing the SLE PtDA
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Lupus Patients
Number analyzed (Participants) | 1828
Participants
  Patient perception of DA Usefulness in decision-making | 1640
  Patient perception of DA Usefulness for information adequacy | 1448

ADVERSE EVENTS:
Time Frame: 6 months
Description: Our evidence-based patient-centered lupus PtDA is an educational tool that addresses important preference-sensitive treatment decisions faced by patients with SLE by providing balanced information.
Arm/Group | Lupus Patients
All-Cause Mortality (participants affected / at risk) | 0/2005
Serious Adverse Events (participants affected / at risk) | 0/2005
Other Adverse Events (participants affected / at risk) | 0/2005

LIMITATIONS AND CAVEATS:
We had few private practice clinics. Most sites were largely academic center clinics. Potential applications of the SLE PtDA to other settings are unexplored to date. Most outcome measures were patient-reported and subjective in nature and therefore may be impacted by social desirability. Satisfaction, acceptability and feasibility, likely had ceiling effects. Not every participant completed all follow-up surveys. Actual sustainability in these clinics cannot be assessed until years have passed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Doc2 (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03735238/Prot_SAP_ICF_000.pdf